CLINICAL TRIAL: NCT00312468
Title: Mechanisms of Atherosclerosis and CVD in HIV+ Women
Brief Title: Examining the Link Between Heart Disease and HIV Infection in Women
Status: Completed | Type: Observational
Sponsor: Albert Einstein College of Medicine (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert Kaplan, Professor of Epidemiology, Albert Einstein College of Medicine
Other Study IDs: 1334; 1R01HL083760 (NIH); 1R01HL126543 (NIH); 1R01HL095140 (NIH)
Record Dates: First submitted 2006-04-06; First posted 2006-04-10 (Estimated); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Cardiovascular Diseases; Atherosclerosis; Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: AIDS
MeSH Terms: conditions — Cardiovascular Diseases; Atherosclerosis; Acquired Immunodeficiency Syndrome; HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
Recent studies have shown that HIV infected individuals have an increased risk of developing heart disease, but the reason for this is not fully understood. This study will examine ultrasound test results of blood vessels and laboratory data of HIV infected and HIV uninfected women to examine the link between heart disease and HIV infection.

DETAILED DESCRIPTION:
HIV infected individuals are at increased risk for developing atherosclerosis, which is a build-up of plaque within the arteries and which may lead to various forms of heart disease. It is unknown, however, why individuals with HIV are more susceptible to heart disease compared to others. Atherosclerosis may develop more rapidly due to HIV infection, the use of antiretroviral medications, or a combination of the two. HIV lipodystrophy syndrome, in which body fat distribution is altered, may also be a risk factor. If heart disease is not properly treated, individuals place themselves at risk for heart attacks, strokes, or organ failure. In previous studies involving HIV and heart disease, women have been under-represented. This study will examine a group of women participating in the Women's Interagency HIV Study (WIHS), which is examining the impact of HIV infection and its clinical, laboratory, and psychosocial effects in women. By using ultrasound imaging, the progression of subclinical atherosclerosis will be assessed. WIHS study data will then be used to examine possible relationships between atherosclerosis and factors associated with HIV infection in women. The results of this study will have major implications for the development of strategies to predict, prevent, or reverse atherosclerosis and heart disease in HIV infected individuals.

This 4-year study will enroll 750 HIV infected women and 250 HIV uninfected women who are participating in the WIHS study. Participants will undergo an initial ultrasound imaging of the neck to measure the size and thickness of the arteries. They will return for a repeat ultrasound at Years 2, 3, and 4 to assess any progression of atherosclerosis. Data from the participants' biannual WIHS study visits, including HIV medication usage, viral load and CD4 test results, and occurrence of AIDS and other illnesses, will be reviewed. Results of participant's inflammation marker tests, which may indicate the presence of atherosclerosis, including white blood cell count, C-reactive protein, E-selectin, and intercellular adhesion molecule 1, will also be reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Women enrolled in the WIHS HIV cohort study

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women enrolled in the WIHS HIV cohort study
Sampling Method: Non-Probability Sample
Enrollment: 1011 (Actual)
Dates: Start 2006-10; Primary Completion 2012-12 (Actual); Study Completion 2012-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Kaplan, PhD, Principal Investigator — Albert Einstein College of Medicine